CLINICAL TRIAL: NCT06745115
Title: Detection of Sepsis Occurrence by Using Blood Fluorescence
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: University of Macau (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-KY133-01
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: blood fluorescence; Sepsis; early detection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
  Interventions: Diagnostic Test: Blood fluorescence metabolite analyzer
- Sepsis Patient Group: Patients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, will be screened and confirmed by a physician to meet the inclusion criteria. After physician confirmation that the inclusion criteria are met, patients will be informed and asked to sign an informed consent form. Blood samples (10 cc) will be collected within 24 hours before and after hospitalization entry. One week post-discharge and on the 28th day post-diagnosis, a nurse will follow up to inquire about their health status.
  Interventions: Diagnostic Test: Blood fluorescence metabolite analyzer
- Infected Non-Sepsis Patient Group: Patients with infections and a SOFA score of 1 will be screened and confirmed by a physician to meet the inclusion criteria. After obtaining informed consent, a nurse will collect a 10 cc blood sample within 24 hours of qualification. Within 7 days of ICU admission, physicians will assess whether patients with non-sepsis infections progress to sepsis. If so, these patients will be categorized into the sepsis patient group.
  Interventions: Diagnostic Test: Blood fluorescence metabolite analyzer

INTERVENTIONS:
Diagnostic Test: Blood fluorescence metabolite analyzer — This study does not involve Intervention. The fluorescence intensity quantified by the blood fluorescence metabolite analyzer does not affect or interfere with clinical diagnosis and treatment. In both the early and late stages of sepsis, a significant increase in inflammatory free radicals changes the optical properties of the patient's blood, distinguishing it from that of healthy individuals. To explore this phenomenon, 10 cc of fasting blood is drawn from patients who pass our screening criteria. This sample is then centrifuged in accordance with our detailed standard operating procedures to ready it for analysis. Subsequently, the fluorescence intensity of the blood is measured quantitatively using a precisely calibrated blood fluorometer, which is specifically designed to detect subtle variations indicative of both early and late sepsis. This entire process is executed under stringent quality control protocols to ensure the reliability and accuracy of the results.

SUMMARY:
This study adopted a case-control study method to explore a reagent-free, highly sensitive, and frequently screened blood fluorescence metabolite analyzer for sepsis, which can detect the emergence of inflammatory free radicals before organ damage and shorten the diagnosis time of sepsis.

DETAILED DESCRIPTION:
Currently, clinical practice lacks an effective screening method for early detection and prediction of sepsis. This gap hinders timely differential diagnosis, leading to severe shock and increased mortality rates. Although the qSOFA score is highly specific, it is not devoid of false negatives. Typically, by the time sepsis is confirmed using the qSOFA (≥ 2) and SOFA (≥ 2) scores as gold standards, the patient may already be suffering from organ damage, thus escalating the risk of death. Early-stage septic patients exhibit a surge in inflammatory free radicals, altering the optical characteristics of their blood compared to that of healthy individuals. Based on this, we hypothesize that a blood fluorometer could detect these early changes in septic patients, enabling rapid and accurate diagnosis to mitigate mortality rates. This study will conduct a case-control investigation, collecting blood from both admitted and discharged patients, with the aim of developing a reagent-free, highly sensitive blood fluorescence metabolite analyzer. This device will be capable of frequent sepsis screenings, detecting inflammatory free radicals before organ damage occurs, thereby reducing the time to sepsis diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
2. Sepsis Experimental Group: Patients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, will be screened and confirmed by a physician to meet the inclusion criteria.
3. Non-septic Severe Control Group: Patients with suspected or confirmed infections, having a SOFA score of 1, will be screened and confirmed by a physician to meet the inclusion criteria.

Exclusion Criteria: minors, pregnant, individuals with mental illnesses, and other vulnerable groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
  2. Sepsis Experimental Group: Inpatients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, will be screened and confirmed by a physician to meet the inclusion criteria.
  3. Non-septic Severe Control Group: Inpatients with suspected or confirmed infections, having a SOFA score of 1, will be screened and confirmed by a physician to meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
specificity and sensitivity of blood fluorescence intensity in diagnosing sepsis. | 1 year
  The primary outcome variable for this clinical trial is the specificity and sensitivity of blood fluorescence intensity in diagnosing sepsis.

SECONDARY OUTCOMES:
The secondary outcome variables consist of correlation coefficients. These coefficients show the relationship between the fluorescence intensity of participants' blood and several other factors, including the length of their hospital stay. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- zhujiang Hospital, Guangzhou, Guangdong, China